CLINICAL TRIAL: NCT04989959
Title: An Exploratory Study of [18F]PT2385 PET/CT in Patients With Renal Cell Carcinoma
Brief Title: [18F]PT2385 PET/CT in Patients With Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Orhan Kemal Oz (Other)
Responsible Party: Sponsor-Investigator, Orhan Kemal Oz, Professor and Division Chief, Department of Radiology, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2021-0592
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pre-Surgical (Experimental): Patients with suspected RCC planned for surgery
  Interventions: Drug: [18F]PT2385; Procedure: Positron Emission Tomography/Computed Tomography
- Metastatic or VHL Syndrome (Experimental): Patients with metastatic ccRCC or VHL syndrome and RCC
  Interventions: Drug: [18F]PT2385; Procedure: Positron Emission Tomography/Computed Tomography; Procedure: Biopsy
- Planned belzutifan treatment (Experimental): Patients with VHL syndrome with RCC, CNS hemangioblastoma, and/or pancreatic neuroendocrine tumor(s) planning to start belzutifan.
  Interventions: Drug: [18F]PT2385; Procedure: Positron Emission Tomography/Computed Tomography

INTERVENTIONS:
Drug: [18F]PT2385 — [18F]PT2385 infusion
Procedure: Positron Emission Tomography/Computed Tomography — PET/CT scan after [18F]PT2385 infusion
  Other Names: PET/CT
Procedure: Biopsy — CT-guided tumor biopsy
  Arms: Metastatic or VHL Syndrome

SUMMARY:
This is an exploratory study to assess [18F]PT2385 Positron Emission Tomography/Computed Tomography (PET/CT) in patients with renal cell carcinoma (RCC). This is an open-label, nontherapeutic trial. The main objective is to correlate hypoxia-inducible factor-2alpha (HIF2α) levels as determined by an investigational [18F]PT2385 PET/CT scan with the levels on subsequently obtained tissue by HIF2α immunohistochemistry (IHC). There will be three cohorts. The first pre-surgical cohort will have [18F]PT2385 PET/CT prior to nephrectomy. The uptake and retention on Positron Emission Tomography (PET), quantified as standardized uptake value (SUV) max and mean, abbreviated SUV henceforth will be correlated with HIF2α levels by IHC on the primary tumor. The second cohort will comprise patients with metastatic clear cell renal carcinoma (ccRCC). SUV will be correlated with HIF2α levels measured by IHC on a biopsy sample from a metastasis. Both low- and high-avidity sites will be biopsied and tracer uptake correlated with HIF2α IHC. A third cohort will include patients with Von Hippel-Lindau (VHL) syndrome and any of the following disease manifestations - RCC, central nervous system (CNS) hemangioblastoma, and/or pancreatic neuroendocrine tumor(s). Investigational imaging will evaluate HIF2α expression within a tumor type and across different tumor types. A biopsy is encouraged but not mandatory for this cohort.

DETAILED DESCRIPTION:
HIF2α is an emerging therapeutic target in RCC. Proof-of-principle experiments in mice have demonstrated the feasibility of PET/CT imaging with novel radiotracers, [11C] and [18F]PT2385, to assess HIF2α expression in RCC. [18F]PT2385 has been proposed in this study for practical imaging of HIF2α.

This is a non-therapeutic research study. Patients with localized or metastatic RCC will undergo imaging with [18F]PT2385. Patients will have the opportunity to ask questions regarding the procedure. A peripheral intravenous line will be placed for [18F]PT2385 administration. Patients will be injected with [18F]PT2385 intravenously and evaluated by PET/CT.

Up to 15 subjects will undergo a dynamic PET scanning and multi-time point whole body imaging to determine the intratumoral tracer kinetics, the optimal time point for whole body imaging, as well as to calculate human dosimetry. In the first 3 subjects, a dynamic scan over the kidneys will be performed for approximately 25 minutes. Upon completion of the dynamic scan, a whole-body scan will be acquired to yield a whole body distribution at approximately 35 minutes. These 3 subjects will be asked to return for delayed whole body images at 120 and 240 minutes post injection. In up to 7 additional subjects, a dynamic scan will be acquired for 55 minutes followed by an immediate whole body scan to yield whole body distribution at approximately 65 minutes. Additional whole-body images will be acquired at 120 and 240 minutes post-injection.

The pre-surgical cohort of 5 subjects will receive one PET/CT scan at the optimal time point determined from the first 15 subjects. Subsequently, surgery will be performed, and SUV from the PET scans will be correlated with HIF2α levels by IHC on the surgical specimen.

A second cohort of 10 subjects with metastatic RCC will be evaluated. Patients with metastatic disease should all have a previous tissue diagnosis, and this cohort will focus on ccRCC patients. Subjects with metastatic ccRCC will be injected with [18F]PT2385 by intravenous (IV) push and will have a whole-body [18F]PT2385 PET/CT at a time considered optimal based on imaging studies performed in cohort 1. A mandatory biopsy will be performed, and up to 4 suitable core tissue samples will be obtained.

A third cohort of 5 subjects with VHL syndrome and any of the following disease manifestations - RCC, CNS hemangioblastoma, and/or pancreatic neuroendocrine tumor(s)- will be evaluated. Subjects will be injected with [18F]PT2385 by IV push and will have a whole-body [18F]PT2385 PET at a time considered optimal based on imaging studies performed in the cohort 1. A biopsy is encouraged but not mandatory. If pursued, the biopsy will be performed in a similar fashion as that performed in cohort 2. Future biopsies per standard of care may be utilized for HIF2α and/or other biomarker analyses.

Following dosimetry studies, a subset of patients may undergo repeat [18F]PT2385 PET studies.

Patients in all cohorts will receive standard or experimental treatment for RCC at the discretion of the treating physician.

Recently available at UTSW, Positron Emission Tomography/Magnetic Resonance Imaging (PET/MRI) may be used instead of PET/CT at the physician/investigator discretion wherever PET/CT is mentioned. PET/MRI is a novel hybrid technology that combines physiologic information from a PET scan and detailed anatomic images from an magnetic resonance imaging (MRI) scan. PET/MRI has the potential to increase imaging quality/diagnostic accuracy while reducing radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent that includes study interventions (PET/CT and, if cohort 2, mandatory biopsy).
* Ability to lie still for a 30- to 60-minute PET/CT scan.
* One of the following:

  1. Cohort 1. Patients with suspected RCC planned for surgery.
  2. Cohort 2. Patients with metastatic ccRCC or VHL syndrome and RCC. Biopsy is required (planned resection for treatment reasons of a metastatic site is acceptable in lieu of the biopsy).
  3. Cohort 3. Patients with VHL syndrome with RCC, CNS hemangioblastoma, and/or pancreatic neuroendocrine tumor(s) planning to start belzutifan.
* Patients with liver dysfunction will be considered "patients of special interest," and enrollment is allowed with or without criteria outlined for Cohorts 1-3. Liver dysfunction is defined clinically and is typically supported by abnormalities in imaging or laboratory studies (alanine / aspartate amino-transferase, bilirubin, alkaline phosphatase, or international normalized range (INR) for prothrombin time).
* Women of child-bearing potential must agree to undergo and have documented a negative pregnancy test on the day of [18F]PT2385 administration. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or celibate by choice) who meets the following criteria:

  1. Has not undergone a hysterectomy or bilateral oophorectomy; or
  2. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

* Uncontrolled severe and irreversible intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Claustrophobia or other contraindications to PET/CT.
* Subjects must not weigh more than the maximum weight limit for the table for the PET/CT scanner where the study is being performed (>200 kilograms or 440 pounds).
* For cohort 2 patients, lack of suitable sites for mandatory biopsy. For example, patients with metastatic disease restricted to the lungs that would require percutaneous biopsies with associated risk of bleeding and pneumothorax will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2027-08-18 (Estimated)

PRIMARY OUTCOMES:
Correlation between [18F]PT2385 and HIF2α | Up to 5 years
  Correlation between [18F]PT2385 PET avidity and HIF2α expression in primary tumors
Correlation between [18F]PT2385 and HIF2α IHC | Up to 5 years
  Correlation between [18F]PT2385 PET avidity and HIF2α expression by IHC

CONTACTS AND LOCATIONS:
Overall Officials: James Brugarolas, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States